CLINICAL TRIAL: NCT00187018
Title: Marrow Mesenchymal Cell Therapy for Osteogenesis Imperfecta: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOD2
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2007-05

CONDITIONS: Osteogenesis Imperfecta
Keywords: Collagen Disease
MeSH Terms: conditions — Osteogenesis Imperfecta; Collagen Diseases | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Bone marrow transplant

SUMMARY:
Osteogenesis imperfecta (OI) is a genetic disease for which there is currently no known cure. OI causes the osteoblasts (bone-forming cells in the body) to grow poorly, which slows the growth of children with the disease and causes their bones to bend and break easily. Some forms of osteogenesis imperfecta may cause severe disability and even death. In previous research studies performed at St. Jude, it was found that children treated with bone marrow transplant (infusion of healthy immature blood-forming cells) began to grow faster, had more minerals (material that helps make the bones strong) in their bones, and broke their bones less often than before the bone marrow transplant. Several months after the bone marrow transplant however, body growth once again began to slow down. In this research study, children with osteogenesis imperfecta will receive another infusion of bone marrow cells but without any chemotherapy. The marrow cells will come from the same bone marrow donor as their previous bone marrow transplant. It is hoped that by removing the CD3+ cells (a type of white blood cells that attack other cells that are not like themselves) from the donated bone marrow, the subject's body will be infused quite safely and that body growth and bone strength will increase. The CD3+ cells will be removed from the donor bone marrow by use of a machine called the CliniMACS System. This machine has not been approved for use in the United States by the Food and Drug Administration (FDA). The use of this device is considered experimental.

ELIGIBILITY:
Inclusion Criteria:

* Must have been previously enrolled on TOIT protocol at St. Jude Children's Research Hospital
* Must have original bone marrow donor available and willing to participate as a donor
* Normal liver function
* Hemoglobin >10gm/dl

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To find out the effects (good and bad) of bone marrow cell infusions using donor bone marrow that has had CD3+ cells removed
To find out if there is any effect on the growth rate of children with osteogenesis imperfecta who receive donor bone marrow which has had CD3+ cells removed
To find out if there is any effect on the total bone mineral content of children with OI
who receive donor bone marrow which has had CD3+ cells removed

SECONDARY OUTCOMES:
To find out the effect of the CD3 washed-out marrow cell therapy on the growth rate of the children

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hale, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Otsuru S, Gordon PL, Shimono K, Jethva R, Marino R, Phillips CL, Hofmann TJ, Veronesi E, Dominici M, Iwamoto M, Horwitz EM. Transplanted bone marrow mononuclear cells and MSCs impart clinical benefit to children with osteogenesis imperfecta through different mechanisms. Blood. 2012 Aug 30;120(9):1933-41. doi: 10.1182/blood-2011-12-400085. Epub 2012 Jul 24. PMID 22829629
- See also: St. Jude Children's Research Hospital — http://www.stjude.org